CLINICAL TRIAL: NCT02766023
Title: Phase II-b Randomized Double-Blind Placebo-Controlled Trial of Lactobacillus Crispatus CTV-05 (LACTIN-V) to Prevent the Recurrence of Bacterial Vaginosis
Brief Title: LACTIN-V Study for Recurrent Bacterial Vaginosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14-0029; HHSN272201300014I
Record Dates: First submitted 2016-04-21; First posted 2016-05-09 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2017-04-05

CONDITIONS: Bacterial Vaginosis
Keywords: CTV-05; LACTIN-V; Lactobacillus; MetroGel®; Vaginitis
MeSH Terms: conditions — Vaginosis, Bacterial; Vaginitis | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LACTIN-V (Experimental): Subjects receive 5-day course of metronidazole gel 7.5 mg/gm daily applied vaginally. Subjects then receive LACTIN-V 2x10^9 cfu/dose applied vaginally for 5 days then twice weekly for 10 weeks. N=152
  Interventions: Biological: Lactobacillus crispatus CTV-05; Drug: Metronidazole
- Placebo (Placebo Comparator): Subjects receive 5-day course of metronidazole gel 7.5 mg/gm daily applied vaginally. Subjects then receive placebo applied vaginally for 5 days then twice weekly for 10 weeks. N=76
  Interventions: Drug: Metronidazole; Other: Placebo

INTERVENTIONS:
Biological: Lactobacillus crispatus CTV-05 — LACTIN-V is an intravaginal live biotherapeutic product composed of Lactobacillus crispatus CTV-05 (LACTIN-V, Osel Inc) in a vaginal applicator. Subjects receive 2x10^9 cfu/dose applied vaginally daily x 5 days then twice weekly x 10 weeks.
  Arms: LACTIN-V
Drug: Metronidazole — Metronidazole is a nitroimidazole. Metronidazole gel (MetroGel) is applied vaginally 7.5 mg/gm daily for 5 days
Other: Placebo — Placebo formulation applied vaginally, daily x 5 days then twice weekly x 10 weeks.
  Arms: Placebo

SUMMARY:
This Phase 2b trial is designed to provide a screening evaluation for the hypothesis that, following a 5-day treatment with MetroGel® to treat BV, L. crispatus CTV-05 (LACTIN-V, Osel, Inc.) administered at 2 x 10^9 cfu/dose using a vaginal applicator reduces the 12-week incidence of BV recurrence when compared to placebo. The primary objectives of this study are: 1) To estimate the efficacy of repeated doses of LACTIN-V (2 x 10^9 cfu/dose) as compared to placebo in preventing BV recurrence by 12 weeks following treatment of BV with MetroGel vaginal gel (MetroGel). 2) To assess the safety of LACTIN-V over 24 weeks by comparing the incidence of AEs between individuals randomized to LACTIN-V or placebo.

DETAILED DESCRIPTION:
This is a Phase II-b multicenter randomized double-blind placebo-controlled trial to assess the efficacy of repeated doses of LACTIN-V compared to placebo in preventing BV recurrence in women diagnosed with BV. The study will also assess the safety of LACTIN-V by comparing the incidence of AEs between women randomized to LACTIN-V or placebo. The study plans to enroll 228 non-pregnant, pre-menopausal women age 18 to 45 years. Women will be randomized 2:1 to receive LACTIN-V or placebo. Potentially eligible women will start a standard 5-day course of MetroGel. Women will return to the study clinic within 2 days after completing the 5-day course of MetroGel to re-evaluate eligibility criteria and review the BV test results from the screening visit. Women with Amsel criteria > /=3 and Nugent score 4-10 will be instructed to administer the LACTIN-V or placebo at home for 5 consecutive days and then twice weekly for 10 weeks. The primary objectives of this study are: 1) To estimate the efficacy of repeated doses of LACTIN-V (2 x109 cfu/dose) as compared to placebo in preventing BV recurrence by 12 weeks following treatment of BV with MetroGel vaginal gel (MetroGel). 2) To assess the safety of LACTIN-V over 24 weeks by comparing the incidence of AEs between individuals randomized to LACTIN-V or placebo. Secondary objectives are: 1) To investigate the colonization of LACTIN-V (presence of L. crispatus CTV-05 in the vaginal specimen) and fluctuations over 12 weeks, in relation to menses and sexual intercourse 2) To evaluate user acceptability and tolerability of LACTIN-V over 12 weeks, including perceptions around method of delivery and dosing. 3) To measure long-term colonization of LACTIN-V at 24 weeks (12 weeks after last dosing) 4) To estimate the long-term efficacy of repeated doses of LACTIN-V (2 x 109 cfu/dose) as compared to placebo in preventing BV recurrence at 24 weeks (12 weeks after last dosing)

ELIGIBILITY:
Inclusion Criteria:

1. Capable of reading and writing English and voluntarily provide written informed consent to participate in the study and comply with all study procedures 2. Untreated BV (asymptomatic or symptomatic) as diagnosed during the screening visit defined by >/=3 Amsel criteria. Note: Amsel criteria include the following: --Homogeneous, thin, grayish-white discharge that smoothly coats the vaginal walls; --Vaginal pH >4.5; --Positive whiff-amine test, defined as the presence of a fishy odor when a drop of 10% potassium hydroxide (KOH) is added to a sample of vaginal discharge; --Presence of clue cells (>20% on microscopy). 3. Untreated BV(asymptomatic or symptomatic) as confirmed in the laboratory using the Nugent scoring system (Nugent Score >/= 4) 4. Otherwise healthy pre-menopausal women 18-45 years of age on the day of screening 5. Regular predictable menstrual cycles or amenorrheic for at least 3 months due to use of a long-acting progestin or continuous use of oral contraceptives 6. Willing to be asked questions about personal medical health and sexual history. 7. Willing to apply study agent vaginally and comply with study examinations. 8. Agree to abstain from sexual intercourse during the first 5 consecutive days of study product administration, 12 hours prior to study visits and for 12 hours after each study product application 9. Agree to abstain from the use of any other intravaginal product throughout the trial period from the time of screening through Visit 7 (Week 24, Day 168) Note: Intravaginal products include contraceptive creams such as Gynol II, gels, foams, sponges, lubricants not approved by the study investigators, and douches. Limit use of tampons during menstruation to unscented products. 10. Must be of non-childbearing potential or if of childbearing potential, must agree to use a reliable method of birth control for the duration of the study Note: Reliable methods of birth control include tubal ligation, male partner with a vasectomy, a steroidal contraceptive (oral, patch, injectable or implantable), IUD, condoms or abstinence.

Exclusion Criteria:

1. Urogenital infection at screening Note: Urogenital infection includes urinary tract infection, Trichomonas (T.) vaginalis, Neisseria (N.) gonorrhoeae, Chlamydia (C.) trachomatis, Treponema (T.) pallidum, or vulvo-vaginal candidiasis. 2. Diagnosis of two or more outbreaks of N. gonorrhoeae, C. trachomatis, T. pallidum, T. vaginalis, or herpes simplex virus (herpes genitalis) within 6 months prior to screening 3. Positive for syphilis or HIV at screening 4. Current pregnancy or within 2 months of last pregnancy and/or currently breastfeeding**. Criteria will be assessed at screening and enrollment. 5. Vaginal or systemic antibiotic or antifungal therapy (other than MetroGel given as part of study procedures) within 21 days of screening or within 30 days of enrollment** 6. Use of disulfiram within past 2 weeks or other contraindication to use of MetroGel** 7. Any condition requiring regular periodic use of systemic antibiotics during participation in the trial 8. Active genital herpes lesion** (if not resolved by enrollment)** 9. Investigational drug use other than LACTIN-V within 30 days or 10 half-lives of the drug, whichever is longer, of enrollment visit** 10. Other planned participation in an investigational drug study while participating in this study** 11. Menopause defined as more than 12 consecutive months of amenorrhea without another known cause including pregnancy 12. IUD insertion or removal, pelvic surgery, cervical cryotherapy or cervical laser treatment within the last 2 months prior to screening 13. Use of vaginal ring (eg, NuvaRing) within 3 days of screening or during the course of the study** 14. Failure to complete 5 days of MetroGel with the last dose taken no later than 48 hours prior to randomization*** 15. Use of new long-acting hormonal treatments. Participant may be enrolled if stable (>3 months) on existing therapy as determined by the principal investigator** 16. Known allergy to any component of LACTIN-V/placebo or MetroGel or to nitroimidazole derivatives or latex (condoms) 17. Any social, medical, or psychiatric condition, including history of drug or alcohol abuse that in the opinion of the investigator would make it unlikely for the participant to comply with the study ** Note: Criteria will be assessed at screening and enrollment. ***Note: Criteria will be assessed at enrollment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California, San Diego - Antiviral Research Center, San Diego, California
  - San Francisco General Hospital - Infectious Diseases, San Francisco, California
  - Cook County Health and Hospitals System - Ruth M Rothstein CORE Center, Chicago, Illinois
  - Washington University School of Medicine in St. Louis - Infectious Disease Clinical Research Unit, St Louis, Missouri

REFERENCES:
- [Derived] Armstrong E, Hemmerling A, Miller S, Burke KE, Newmann SJ, Morris SR, Reno H, Huibner S, Kulikova M, Liu R, Crawford ED, Castaneda GR, Nagelkerke N, Coburn B, Cohen CR, Kaul R. Metronidazole treatment rapidly reduces genital inflammation through effects on bacterial vaginosis-associated bacteria rather than lactobacilli. J Clin Invest. 2022 Mar 15;132(6):e152930. doi: 10.1172/JCI152930. PMID 35113809
- [Derived] Cohen CR, Wierzbicki MR, French AL, Morris S, Newmann S, Reno H, Green L, Miller S, Powell J, Parks T, Hemmerling A. Randomized Trial of Lactin-V to Prevent Recurrence of Bacterial Vaginosis. N Engl J Med. 2020 May 14;382(20):1906-1915. doi: 10.1056/NEJMoa1915254. PMID 32402161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were non-pregnant females with untreated bacterial vaginosis recruited from the clinics conducting the study and from other clinical providers coordinating referrals of eligible women to the study centers. Participants were enrolled between 03JUN2016 and 27AUG2018.
Groups:
- LACTIN-V: Participants receive 5-day course of metronidazole gel 7.5 mg/gm daily applied vaginally. Participants then receive LACTIN-V 2x10^9 cfu/dose applied vaginally for 5 days then twice weekly for 10 weeks. N=152
  Lactobacillus crispatus CTV-05: LACTIN-V is an intravaginal live biotherapeutic product composed of Lactobacillus crispatus CTV-05 (LACTIN-V, Osel Inc) in a vaginal applicator. Participants receive 2x10^9 cfu/dose applied vaginally daily x 5 days then twice weekly x 10 weeks.
  Metronidazole: Metronidazole is a nitroimidazole. Metronidazole gel (MetroGel) is applied vaginally 7.5 mg/gm daily for 5 days
- Placebo: Participants receive 5-day course of metronidazole gel 7.5 mg/gm daily applied vaginally. Participants then receive placebo applied vaginally for 5 days then twice weekly for 10 weeks. N=76
  Metronidazole: Metronidazole is a nitroimidazole. Metronidazole gel (MetroGel) is applied vaginally 7.5 mg/gm daily for 5 days
  Placebo: Placebo formulation applied vaginally, daily x 5 days then twice weekly x 10 weeks.
Period: Overall Study
Arm/Group | LACTIN-V | Placebo
Started | 152 | 76
Completed | 122 | 59
Not Completed | 30 | 17
Not completed — Lost to Follow-up | 23 | 11
Not completed — Pregnancy | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Not Eligible at Enrollment | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all subjects enrolled and randomized into the study.
Groups:
- LACTIN-V: 5-day course of metronidazole gel 7.5 mg/gm daily applied vaginally, then LACTIN-V 2x10^9 cfu/dose applied vaginally for 5 days then twice weekly for 10 weeks.
- Placebo: 5-day course of metronidazole gel 7.5 mg/gm daily applied vaginally, then placebo applied vaginally for 5 days then twice weekly for 10 weeks.
- Total: Total of all reporting groups
Arm/Group | LACTIN-V | Placebo | Total
Number analyzed (Participants) | 152 | 76 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 152 | 76 | 228
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (6.8) | 31.4 (7.1) | 30.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 76 | 228
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 15 | 45
  Not Hispanic or Latino | 122 | 61 | 183
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 64 | 31 | 95
  White | 55 | 26 | 81
  More than one race | 10 | 7 | 17
  Unknown or Not Reported | 14 | 8 | 22
Region of Enrollment [Number; unit: participants]
  United States | 152 | 76 | 228

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants Reporting Product-related Adverse Events (AEs) and Serious Adverse Events (SAEs) in Each Study Arm.
Description: Adverse events and serious adverse events were collected during the entire study period. Relatedness to study product was assessed by the site investigator according to the protocol definition of related as "There is a reasonable possibility that the study product caused the AE. Reasonable possibility means that there is evidence to suggest a causal relationship between the study product and the AE."
Time Frame: Day 1 to Day 168
Population: The safety population included all participants receiving study product. One participant randomized to LACTIN-V was not treated.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 151 | 76
proportion of participants | 0.11 [0.06 to 0.16] | 0.07 [0.03 to 0.15]
Statistical Analysis 1: Comparison: LACTIN-V vs Placebo; Test type: Superiority; p = 0.467, Fisher Exact; Risk Difference (RD) = 0.04, 95% CI 2-sided [-0.10 to 0.18]

2. Primary Outcome: The Proportion of Participants With a Positive BV Diagnosis in Each Study Arm.
Description: A positive BV diagnosis was defined by meeting at least 3 of the 4 Amsel criteria and a Nugent score of 4-10. Amsel criteria are: homogeneous, thin, grayish-white discharge that smoothly coats the vaginal walls; vaginal pH >4.5; positive whiff-amine test, defined as the presence of a fishy odor when a drop of 10% potassium hydroxide is added to a sample of vaginal discharge; and presence of clue cells (>20%) on microscopy. The Amsel score ranges from 0-4, where higher scores mean a worse outcome. The Nugent score is calculated by assessing for the presence of large Gram-positive rods scored as 0 to 4, small Gram-variable rods scored as 0 to 4, and curved Gram-variable rods scored as 0 to 2, and adding all component scores. The Nugent score ranges from 0-10, where higher scores mean a worse outcome. All BV diagnoses following 15 days after enrollment (22 days after commencement of MetroGel treatment) were considered a recurrent episode.
Time Frame: Day 1 to Day 84
Population: The analysis population was the intent-to-treat population (all randomized participants). Missing BV recurrence data was imputed using Last Observation Carried Forward
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 152 | 76
proportion of participants | 0.30 [0.24 to 0.38] | 0.45 [0.34 to 0.56]
Statistical Analysis 1: Comparison: LACTIN-V vs Placebo; Test type: Superiority; p = 0.031, Chi-squared; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.30 to 0.95]

3. Secondary Outcome: The Proportion of Participants Who Are Compliant With the Complete Dose Regimen as Assessed by Participant Reporting and Applicator Staining.
Description: A subject was considered compliant with the assigned study product if she took 4 of the first 5 daily doses and at least 75% of the scheduled doses overall prior to the first diagnosis of BV or through Week 12, whichever occurred first. Compliance was assessed by subject report via the memory aid and, separately, applicator staining of the returned kit. Compliance was assessed on a weekly basis and the time (week) at which the subject became non-compliant was determined by blinded PI review.
Time Frame: Day 1 to Day 84
Population: The analysis population was the intent-to-treat population (all randomized participants).
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 152 | 76
proportion of participants
  Self-report | 0.80 [0.73 to 0.86] | 0.78 [0.67 to 0.86]
  Staining | 0.77 [0.70 to 0.83] | 0.72 [0.61 to 0.81]
Statistical Analysis 1: Comparison: LACTIN-V vs Placebo; Analysis is for self-reported compliance; Test type: Superiority; p = 0.643, Chi-squared; Risk Difference (RD) = 0.03, 95% CI 2-sided [-0.08 to 0.15]
Statistical Analysis 2: Comparison: LACTIN-V vs Placebo; Analysis is for compliance assessed by staining; Test type: Superiority; p = 0.446, Chi-squared; Risk Difference (RD) = 0.05, 95% CI 2-sided [-0.07 to 0.17]

4. Secondary Outcome: Acceptability of LACTIN-V and the Applicator Measured by Self-administered Questionnaires About Acceptability - Categorical Variables on Likert Scale
Description: Participants answered a detailed self-administered questionnaire at Week 12 assessing the acceptability of the study product and the applicator. Questionnaire items included rating aspects of the product and applicator by Likert-scale responses of strongly agree, agree, neutral, disagree and strongly disagree.
Time Frame: Day 84
Population: The analysis population includes all treated participants who completed the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 130 | 63
Participants
  I was satisfied overall with vaginal applicator: Strongly agree | 59 | 22
  I was satisfied overall with vaginal applicator: Agree | 55 | 30
  I was satisfied overall with vaginal applicator: Neutral | 12 | 7
  I was satisfied overall with vaginal applicator: Disagree | 3 | 4
  I was satisfied overall with vaginal applicator: Strongly disagree | 1 | 0
  Satisfied with comfort of vaginal applicator: Strongly agree | 55 | 23
  Satisfied with comfort of vaginal applicator: Agree | 56 | 32
  Satisfied with comfort of vaginal applicator: Neutral | 17 | 5
  Satisfied with comfort of vaginal applicator: Disagree | 1 | 2
  Satisfied with comfort of vaginal applicator: Strongly disagree | 1 | 1
  Satisfied with ease of use of vaginal applicator: Strongly agree | 63 | 31
  Satisfied with ease of use of vaginal applicator: Agree | 58 | 28
  Satisfied with ease of use of vaginal applicator: Neutral | 8 | 2
  Satisfied with ease of use of vaginal applicator: Disagree | 1 | 2
  Satisfied with ease of use of vaginal applicator: Strongly disagree | 0 | 0
  Vaginal health improved with study participation: Strongly agree | 46 | 18
  Vaginal health improved with study participation: Agree | 45 | 18
  Vaginal health improved with study participation: Neutral | 25 | 21
  Vaginal health improved with study participation: Disagree | 10 | 5
  Vaginal health improved with study participation: Strongly disagree | 4 | 1
  Important I use product without partner knowing: Strongly agree | 32 | 12
  Important I use product without partner knowing: Agree | 29 | 15
  Important I use product without partner knowing: Neutral | 45 | 22
  Important I use product without partner knowing: Disagree | 15 | 8
  Important I use product without partner knowing: Strongly disagree | 9 | 6
  Important for me that partner approved of product: Strongly agree | 10 | 6
  Important for me that partner approved of product: Agree | 22 | 10
  Important for me that partner approved of product: Neutral | 34 | 23
  Important for me that partner approved of product: Disagree | 34 | 13
  Important for me that partner approved of product: Strongly disagree | 30 | 11
  I would use the product again: Strongly agree | 72 | 28
  I would use the product again: Agree | 39 | 24
  I would use the product again: Neutral | 11 | 7
  I would use the product again: Disagree | 4 | 3
  I would use the product again: Strongly disagree | 4 | 1

5. Secondary Outcome: Acceptability of LACTIN-V and the Applicator Measured by Self-administered Questionnaires About Acceptability - Likelihood to Use
Description: Participants answered a detailed self-administered questionnaire at Week 12 assessing the acceptability of the study product and the applicator. Questionnaire items included rating aspects of the product and applicator by various measures, including the question, "If a non-antibiotic, clinically proven lactobacillus product were available for treatment and prevention of BV, what are the chances that you would use it?"
Time Frame: Day 84
Population: The analysis population includes all treated participants who completed the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 130 | 63
Participants
  Certain; almost certain | 83 | 37
  Very probable | 25 | 16
  Good possibility | 14 | 7
  Slight possibility | 8 | 2
  No chance; almost no chance | 0 | 1

6. Secondary Outcome: Acceptability of LACTIN-V and the Applicator Measured by Self-administered Questionnaires About Acceptability - Current Partner's Reaction to the Product
Description: Participants answered a detailed self-administered questionnaire at Week 12 assessing the acceptability of the study product and the applicator. Questionnaire items included rating aspects of the product and applicator by various measures, including "My current partner's reaction to the product was..." with the options as listed below.
Time Frame: Day 84
Population: The analysis population includes all treated participants who completed the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 130 | 63
Participants
  Currently does not have a partner | 21 | 10
  Positive | 39 | 23
  Neutral | 31 | 16
  Negative | 9 | 2
  Partner was unaware of product use | 20 | 9
  Unknown | 10 | 3

7. Secondary Outcome: Acceptability of LACTIN-V and the Applicator Measured by Self-administered Questionnaires About Acceptability - Current Partner's Reaction as Influence
Description: Participants answered a detailed self-administered questionnaire at Week 12 assessing the acceptability of the study product and the applicator. Questionnaire items included rating aspects of the product and applicator by various measures, including if their current partner's reaction to the product influenced their use of the product.
Time Frame: Day 84
Population: The analysis population includes all treated participants who completed the questionnaire and had a current partner.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 109 | 53
Participants
  No | 73 | 36
  Yes, and was more likely to use it | 19 | 9
  Yes, and was less likely to use it | 2 | 0
  Unknown | 15 | 8

8. Secondary Outcome: Acceptability of LACTIN-V and the Applicator Measured by Self-administered Questionnaires About Acceptability - Experience Side Effects
Description: Participants answered a detailed self-administered questionnaire at Week 12 assessing the acceptability of the study product and the applicator. Questionnaire items included rating aspects of the product and applicator by various measures, including a Yes/No question about experiencing side effects.
Time Frame: Day 84
Population: The analysis population includes all treated participants who completed the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 130 | 63
Participants
  No | 81 | 44
  Yes | 49 | 19

9. Secondary Outcome: Acceptability of LACTIN-V and the Applicator Measured by Self-administered Questionnaires About Acceptability - Experience of Side Effects Make Less Likely to Use
Description: Participants answered a detailed self-administered questionnaire at Week 12 assessing the acceptability of the study product and the applicator. Questionnaire items included rating aspects of the product and applicator by various measures, including a Yes/No question about experiencing side effects. For those participants who answered Yes to experiencing side effects, a follow-up question asked "would these side effects make you less likely to use the product again?"
Time Frame: Day 84
Population: The analysis population is limited to those participants who answered "Yes" to the question "Did you experience any side effects using the product?"
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 49 | 19
Participants
  Strongly agree | 2 | 1
  Agree | 6 | 3
  Neutral | 7 | 7
  Disagree | 20 | 4
  Strongly disagree | 14 | 4

10. Secondary Outcome: Acceptability of LACTIN-V and the Applicator Measured by Self-administered Questionnaires About Acceptability - Continuous/Discrete Response Regarding Product
Description: Participants answered a detailed self-administered questionnaire at Week 12 assessing the acceptability of the study product and the applicator. Questionnaire items included rating aspects of the product and applicator by various measures, including by rating factors on a 0-10 scale, with 0 being "not at all" and 10 being "extremely".
Time Frame: Day 84
Population: The analysis population includes all treated participants who completed the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 130 | 63
units on a scale
  Effectiveness | 7.53 (2.81) | 6.72 (2.97)
  Comfort | 8.16 (2.22) | 8.07 (2.10)
  Ease of use | 8.99 (1.57) | 8.75 (1.75)
  Vaginal health | 7.37 (2.83) | 7.01 (2.88)
  Other Finding | 8.21 (2.58) | 9.27 (0.64)

11. Secondary Outcome: Acceptability of LACTIN-V and the Applicator Measured by Self-administered Questionnaires About Acceptability - Continuous/Discrete Response Regarding Product Use
Description: Participants answered a detailed self-administered questionnaire at Week 12 assessing the acceptability of the study product and the applicator. Questionnaire items included rating aspects of the product and applicator by various measures, including by rating factors on use of the product on a 0-10 scale, with 0 being "not at all" and 10 being "extremely so".
Time Frame: Day 84
Population: The analysis population includes all treated participants who completed the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 130 | 63
units on a scale
  High frequency | 2.97 (3.20) | 2.63 (3.09)
  Vaginal Dryness | 1.71 (2.66) | 1.37 (2.43)
  Discomfort | 1.53 (2.43) | 1.01 (1.80)
  Messiness | 2.10 (2.82) | 1.68 (2.65)
  Disapproval | 0.98 (2.07) | 0.79 (1.84)
  Other issue | 7.08 (1.69) | 7.62 (1.68)

12. Secondary Outcome: The Proportion of Participants Experiencing Successful Colonization With L. Crispatus CTV-05 Following Dose of Study Product in the LACTIN-V Arm Overall.
Description: Colonization of L. crispatus was determined from the concentrations of L. crispatus species and L. crispatus CTV-05 obtained from qPCR. Successful colonization was defined as: If CTV-05 concentration was above the lower limit of detection (LLOD) and the L. crispatus was above the LLOD, then successful colonization had occurred. If either CTV-05 or L. crispatus concentration was below LLOD or indeterminate, then successful colonization had not occurred. The LLOD for CTV-05 was 660 copies/mL and the LLOD for L. crispatus was 953 copies/mL
Time Frame: Day 1 to Day 84
Population: The analysis population is intent to treat.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 152 | 76
percentage of participants | 0.85 [0.78 to 0.90] | 0.07 [0.03 to 0.14]
Statistical Analysis 1: Comparison: LACTIN-V vs Placebo; Test type: Superiority; p < 0.001, Chi-squared; Odds Ratio (OR) = 79.64, 95% CI 2-sided [29.02 to 218.57]

13. Secondary Outcome: The Proportion of Participants Experiencing Successful Colonization With L. Crispatus CTV-05 Following Dose of Study Product by Occurrence of Intercourse.
Description: as for outcome 12
Time Frame: Day 1
Population: The analysis population includes participants with results at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 149 | 75
Participants
  Condom-less sex acts since last visit: number analyzed (Participants) | 11 | 12
  Condom-less sex acts since last visit | 0 | 0
  No condom-less sex acts since last visit: number analyzed (Participants) | 138 | 63
  No condom-less sex acts since last visit | 4 | 0

14. Secondary Outcome: The Proportion of Participants Experiencing Successful Colonization With L. Crispatus CTV-05 Following Dose of Study Product by Occurrence of Intercourse.
Description: as for outcome 12
Time Frame: Day 28
Population: The analysis population includes participants with results at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 134 | 64
Participants
  Condom-less sex acts since last visit: number analyzed (Participants) | 43 | 26
  Condom-less sex acts since last visit | 37 | 1
  No condom-less sex acts since last visit: number analyzed (Participants) | 91 | 38
  No condom-less sex acts since last visit | 76 | 3

15. Secondary Outcome: The Proportion of Participants Experiencing Successful Colonization With L. Crispatus CTV-05 Following Dose of Study Product by Occurrence of Intercourse.
Description: as for outcome 12
Time Frame: Day 56
Population: The analysis population includes participants with results at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 127 | 58
Participants
  Condom-less sex acts since last visit: number analyzed (Participants) | 39 | 24
  Condom-less sex acts since last visit | 28 | 0
  No condom-less sex acts since last visit: number analyzed (Participants) | 88 | 34
  No condom-less sex acts since last visit | 78 | 1

16. Secondary Outcome: The Proportion of Participants Experiencing Successful Colonization With L. Crispatus CTV-05 Following Dose of Study Product by Occurrence of Intercourse.
Description: as for outcome 12
Time Frame: Day 84
Population: The analysis population includes participants with results at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 131 | 63
Participants
  Condom-less sex acts since last visit: number analyzed (Participants) | 49 | 23
  Condom-less sex acts since last visit | 38 | 0
  No condom-less sex acts since last visit: number analyzed (Participants) | 82 | 40
  No condom-less sex acts since last visit | 64 | 2

17. Secondary Outcome: The Proportion of Participants Experiencing Successful Colonization With L. Crispatus CTV-05 Following Dose of Study Product by Occurrence of Menses.
Description: as for outcome 12
Time Frame: Day 28
Population: The analysis population includes participants with results at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 134 | 64
Participants
  Menses since last visit: number analyzed (Participants) | 109 | 51
  Menses since last visit | 93 | 3
  No menses since last visit: number analyzed (Participants) | 25 | 13
  No menses since last visit | 20 | 1

18. Secondary Outcome: The Proportion of Participants Experiencing Successful Colonization With L. Crispatus CTV-05 Following Dose of Study Product by Occurrence of Menses.
Description: as for outcome 12
Time Frame: Day 56
Population: The analysis population includes participants with results at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 127 | 58
Participants
  Menses since last visit: number analyzed (Participants) | 92 | 44
  Menses since last visit | 76 | 1
  No menses since last visit: number analyzed (Participants) | 35 | 14
  No menses since last visit | 30 | 0

19. Secondary Outcome: The Proportion of Participants Experiencing Successful Colonization With L. Crispatus CTV-05 Following Dose of Study Product by Occurrence of Menses.
Description: as for outcome 12
Time Frame: Day 84
Population: The analysis population includes participants with results at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 131 | 63
Participants
  Menses since last visit: number analyzed (Participants) | 98 | 48
  Menses since last visit | 74 | 2
  No menses since last visit: number analyzed (Participants) | 33 | 15
  No menses since last visit | 28 | 0

20. Secondary Outcome: The Proportion of Participants Experiencing Successful Colonization With L. Crispatus CTV-05 Following Dose of Study Product Overall.
Description: as for outcome 12
Time Frame: Day 1 to Day 168
Population: The analysis population was the intent-to-treat population (all randomized participants).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 152 | 76
percentage of participants | 0.86 [0.80 to 0.91] | 0.08 [0.04 to 0.16]
Statistical Analysis 1: Comparison: LACTIN-V vs Placebo; Test type: Superiority; p < 0.001, Chi-squared; Odds Ratio (OR) = 72.78, 95% CI 2-sided [28.07 to 188.66]

21. Secondary Outcome: The Proportion of Participants With a Positive BV Diagnosis in Each Study Arm.
Description: A positive BV diagnosis was defined by at least 3 of the 4 Amsel criteria and a Nugent score of 4-10. Amsel criteria are: homogeneous, thin, grayish-white discharge that smoothly coats the vaginal walls; vaginal pH >4.5; positive whiff-amine test, defined as the presence of a fishy odor when a drop of 10% potassium hydroxide is added to a sample of vaginal discharge; and presence of clue cells (>20%) on microscopy. The Nugent score is calculated by assessing for the presence of large Gram-positive rods scored as 0 to 4, small Gram-variable rods scored as 0 to 4, and curved Gram-variable rods scored as 0 to 2. All BV diagnoses following 15 days after enrollment (22 days after commencement of MetroGel treatment) were considered a recurrent episode.
Time Frame: Day 1 to Day 168
Population: The analysis population was the intent-to-treat population (all randomized participants).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 152 | 76
percentage of participants | 0.39 [0.31 to 0.47] | 0.54 [0.43 to 0.65]
Statistical Analysis 1: Comparison: LACTIN-V vs Placebo; Test type: Superiority; p = 0.030, Chi-squared; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.31 to 0.94]

22. Secondary Outcome: The Number of Participants Who Discontinued Study Product Early in Each Study Arm Due to Adverse Events.
Description: Tolerability of LACTIN-V and the applicator was measured by the proportion of participants who discontinued the study product prior to completing the dose schedule due to an adverse event.
Time Frame: Day 1 to Day 84
Population: The analysis population included all treated participants. One participant randomized to LACTIN-V was not treated.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 151 | 76
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected through Study Week 24.
Description: For events solicited on a Memory Aid, a participant was considered to have an event if it was reported as experienced at any time during the memory aid period.
Arm/Group | LACTIN-V | Placebo
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/76
Serious Adverse Events (participants affected / at risk) | 1/151 | 0/76
Other Adverse Events (participants affected / at risk) | 131/151 | 60/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LACTIN-V (N=151) | Placebo (N=76)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LACTIN-V (N=151) | Placebo (N=76)
Vulvovaginal candidiasis (Infections and infestations) | 14 (16) | 3 (3)
Vulvovaginal mycotic infection (Infections and infestations) | 11 (15) | 5 (5)
Hypertension (Vascular disorders) | 11 (12) | 4 (4)
Vaginal haemorrhage (Reproductive system and breast disorders) | 38 (38) | 22 (22) — Solicited as "Vaginal bleeding other than menstruation"
Vaginal discharge (Reproductive system and breast disorders) | 95 (95) | 46 (46) — Solicited as "Abnormal vaginal discharge"
Vaginal odour (Reproductive system and breast disorders) | 80 (80) | 34 (34) — Solicited as "Abnormal vaginal odor"
Pruritus genital (Reproductive system and breast disorders) | 87 (87) | 34 (34) — Solicited as "Genital itching"
Genital discomfort (Reproductive system and breast disorders) | 48 (48) | 19 (19) — Solicited as "Genital burning"
Genital discomfort (Reproductive system and breast disorders) | 62 (62) | 20 (20) — Solicited as "External genital irritation"
Genital swelling (Reproductive system and breast disorders) | 30 (30) | 10 (10) — Solicited as "External genital swelling"
Genital rash (Reproductive system and breast disorders) | 21 (21) | 7 (7) — Solicited as "Genital rash"
Nausea (Gastrointestinal disorders) | 26 (26) | 8 (8)
Vomiting (Gastrointestinal disorders) | 15 (15) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 59 (59) | 27 (27) — Solicited as "Abdominal pain/cramps"
Diarrhea (Gastrointestinal disorders) | 31 (31) | 12 (12)
Constipation (Gastrointestinal disorders) | 34 (34) | 6 (6)
Dysuria (Renal and urinary disorders) | 29 (29) | 8 (8) — Solicited as "Pain/burning with urination"
Pollakiuria (Renal and urinary disorders) | 36 (36) | 13 (13)
Headache (Nervous system disorders) | 48 (48) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT02766023/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT02766023/SAP_001.pdf